CLINICAL TRIAL: NCT01957462
Title: Investigation of Two Newly Developed 1-piece Convex Baseplates in Subjects With Ileostomy and Colostomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Coloplast A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: CP239
Record Dates: First submitted 2013-08-06; First posted 2013-10-08 (Estimated); Results first posted 2014-08-11 (Estimated); Last update posted 2016-09-26 (Estimated); Status verified 2016-08

CONDITIONS: Ileostomy - Stoma; Colostomy - Stoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- FirstColplast Test V, Then Coloplast Test X (Experimental): The subject tests two experimental coloplast products in a randomised order. Coloplast Test product V and after cross over ColoplastTest product X
  Interventions: Device: Coloplast Test V; Device: Coloplast Test X
- First Coloplast Test X, Then Coloplast Test V (Experimental): The subjects test the two experimental Coloplast products in a randomised order: Coloplast Test product X and after cross over Coloplast Test product V
  Interventions: Device: Coloplast Test V; Device: Coloplast Test X

INTERVENTIONS:
Device: Coloplast Test V — Coloplast Test product V is a newly developed 1-piece ostomy appliance
  Other Names: Coloplast 1-piece convex Test product V
Device: Coloplast Test X — Coloplast Test X is a newly developed 1-piece ostomy appliance
  Other Names: Coloplast 1-piece convex Test product X

SUMMARY:
The aim of the current investigation is to develop new soft and more flexible 1-piece convex ostomy products.

ELIGIBILITY:
Inclusion Criteria:

1. Have given written informed consent and signed letter of authority.
2. Are at least 18 years of age and have full legal capacity.
3. Have had their ostomy (ileo- or colostomy) for at least 3 months.
4. Have used a 1-piece convex ostomy product during the last month.
5. Are willing and able to comply with investigation procedures.
6. Have a ostomy with a diameter of 33 mm or less.

Exclusion Criteria:

1. Currently suffering from peristomal skin problems (i.e. bleeding or broken skin).
2. Currently receiving or have within the past 2 month received radio- and/or chemotherapy.
3. Currently receiving or have within the past month received local (peristomal area) or systemic steroid treatment.
4. Are pregnant or breastfeeding.
5. Have a loop ostomy (also called double-barrel or ostomy with two outlets).
6. Known hypersensitivity toward any of the test products.
7. Use irrigation during the investigation (flush the stoma with water).
8. Participating in other interventional clinical investigations or have previously participated in this investigation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2013-04; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Birte P Jakobsen, MD, Principal Investigator — Coloplast A/S
Locations (1):
- Coloplast A/S, Humlebæk, Denmark

RESULTS

PARTICIPANT FLOW:
Period: Test Period 1
Arm/Group | FirstColplast Test V, Then Coloplast Test X | First Coloplast Test X, Then Coloplast Test V
Started | 16 | 15
Completed | 14 | 15
Not Completed | 2 | 0
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Adverse Event | 1 | 0
Period: Test Period 2
Arm/Group | FirstColplast Test V, Then Coloplast Test X | First Coloplast Test X, Then Coloplast Test V
Started | 14 | 15
Completed | 14 | 15
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Arm/Group | All Subjects
Number analyzed (Participants) | 31
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.4 (12.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24
  Male | 7

OUTCOME MEASURES:

1. Primary Outcome: Degree of Leakage
Description: The degree of leakage is measured using a 32-point scale developed by Coloplast A/S, where 0 represents No leakage (the best possible outcome) and 32 points represents full plate leakage (worst possible outcome).
  The degree of leakage is measured at each baseplate change
Time Frame: 14 days
Measure: Mean (Standard Deviation); unit: units on a scale
Units Other Than Participants: baseplates
Groups:
- Test V: The results presented for the subjects testing Coloplast Test V
- Test X: the results presented for the subjects testing Test X
Arm/Group | Test V | Test X
Number analyzed (Participants) | 31 | 29
Number analyzed (baseplates) | 357 | 336
units on a scale | 3.5 (5.0) | 3.1 (5.1)

ADVERSE EVENTS:
Time Frame: 28+/- 3 days
Arm/Group | Test V | Test X
Serious Adverse Events (participants affected / at risk) | 1/31 | 1/29
Other Adverse Events (participants affected / at risk) | 13/31 | 13/29
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Test V (N=31) | Test X (N=29)
constipation (Gastrointestinal disorders) | 0 (0) | 1 (1) — Not related to device
Absess in the bowl ( by a fistel channel 2 mm from stoma) (Gastrointestinal disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Test V (N=31) | Test X (N=29)
peristomal skin irritation (Skin and subcutaneous tissue disorders) | 7 (8) | 7 (12) — related to device ( AE categorised ad unlikely-, possibly-, probably--and definitely- related are defined as related AEs)
Peristomal Itching (Skin and subcutaneous tissue disorders) | 5 (8) | 1 (1) — related to the device
Peristomal skin Pain (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
broken skin (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Petekkie/pressure mark (peristomal) (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (4) — related to device
Pain and sorness by stoma and´in bowl (Gastrointestinal disorders) | 1 (1) | 0 (0) — Not related to device
Obstipation (Gastrointestinal disorders) | 0 (0) | 1 (1) — Not related to device
dehydration due to obstpation (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
fatigue (General disorders) | 0 (0) | 1 (1)
Pain in bowl (Gastrointestinal disorders) | 1 (1) | 0 (0) — not related to device
Diarrhea (Gastrointestinal disorders) | 1 (1) | 0 (0) — not related to device
Nausea (General disorders) | 1 (1) | 0 (0) — not related to device
sore throat (Infections and infestations) | 0 (0) | 1 (1) — not related to device

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes